CLINICAL TRIAL: NCT02812251
Title: A Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-61393215 in Healthy Subjects
Brief Title: Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-61393215 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108182; 61393215EDI1001 (Other: Janssen-Cilag International NV); 2016-000822-20 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-06-24 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (10):
- Part 1: Cohort 1 (Experimental): Participants will receive 1 milligram (mg) JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 2 (Experimental): Participants will receive 5 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 3 (Experimental): Participants will receive 15 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 4 (Experimental): Participants will receive 30 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 5 (Experimental): Participants will receive 45 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 6 (Experimental): Participants will receive 60 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 7 (Experimental): Participants will receive 90 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1: Cohort 8 (Experimental): Participants will receive 120 mg JNJ-61393215 or placebo.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 2 (Experimental): Participants will receive JNJ-61393215 (dose to be determined).
  Interventions: Drug: JNJ-61393215
- Part 3 (Experimental): Participants will receive JNJ-61393125 (dose to be determined) or placebo under fed conditions.
  Interventions: Drug: JNJ-61393215; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-61393215 — JNJ-61393215 (projected dose levels as described above for Part 1) will be administered as an oral suspension.
Drug: Placebo — Matching placebo will be administered.
  Arms: Part 1: Cohort 1; Part 1: Cohort 2; Part 1: Cohort 3; Part 1: Cohort 4; Part 1: Cohort 5; Part 1: Cohort 6; Part 1: Cohort 7; Part 1: Cohort 8; Part 3

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of JNJ-61393215 versus placebo after single oral dose administration under fasted (ascending dose levels) and fed condition, to characterize the pharmacokinetics of JNJ-61393125 in plasma, cerebrospinal fluid (CSF) and urine after single oral dose administration and to investigate the effect of food (high fat/high calorie) on the pharmacokinetics of JNJ-61393215 following single oral dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI) between 18 and 30 kilogram per meter square kg/m^2, inclusive (BMI = weight/height^2)
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening and admission to the clinical unit. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable. The presence of Left Bundle Branch Block (LBBB), Atrioventricular (AV) Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD] will lead to exclusion
* Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology or urinalysis are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities to be not clinically significant
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository during the study and for 3 months after receiving the last dose of study drug. All men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partner should also use an appropriate method of birth control for at least the same duration.
* Healthy male participants between 18 and 54 years of age, inclusive for Part 1 and 3
* Healthy male and female participants between 55 and 75 years of age, inclusive in Part 2

Exclusion Criteria:

* Participant has a history of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic (including coagulation disorders), rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness. Minor deviations, which are not considered to be of clinical significance to both the investigator and to the Janssen Safety Responsible Physician, are acceptable
* Participant has estimated glomerular filtration rate (eGFR) less than (<) 60 milliliters per minute per 1.73 meter square (mL/min/1.73m^2) at Screening
* Participant has a heart rate less than (<) 50 beats per minute (bpm) at Screening or at admission to the clinical unit
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* Participant has Left Bundle Branch Block (LBBB), Atrioventricular (AV) Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD]

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events and Serious Adverse Events as a Measure of Safety and Tolerability | Up to follow-up phase (7 to 14 days after study drug administration)
Maximum Plasma Concentration (Cmax) of JNJ-61393125 | Up to Day 4
  The Cmax is the maximum observed plasma concentration.
Last Quantifiable Plasma Concentration (Clast) of JNJ-61393125 | Up to Day 4
  The Clast is the last quantifiable plasma concentration.
Time to Reach Maximum Plasma Concentration (Tmax) of JNJ-61393125 | Up to Day 4
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time of the Last Quantifiable Plasma Concentration (Tlast) of JNJ-61393125 | Up to Day 4
  The Tlast is defined as the time of the last quantifiable plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration of JNJ-61393125 | Up to Day 4
  The (AUC [0-last]) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-61393125 | Up to Day 4
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentrations; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
First Order Rate Constant (Lambda[z]) of JNJ-61393125 | Up to Day 4
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-life (t1/2) of JNJ-61393125 | Up to Day 4
  Elimination half-life (t [1/2]) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Total Clearance (CL/F) of JNJ-61393125 | Up to Day 4
  Total clearance of drug after extravascular administration, uncorrected for absolute bioavailability, calculated as: D/AUC infinity.
Creatinine Clearance (CLcr) of JNJ-61393125 | Up to Day 4

SECONDARY OUTCOMES:
Change From Baseline in NeuroCart test battery Score | Up to Day 2
  Effects of JNJ-61393215 on alertness/sedation will be assessed by means of the NeuroCart test battery (including pharmaco-electroencephalogram [EEG], saccadic eye movements, smooth pursuit, adaptive tracking, body sway, Bond & Lader Visual Analogue Scale (VAS), Bowdle VAS, Swiss Narcolepsy Scale [SNS]).
Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT Fatigue) | Up to Day 2
  The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The total FACIT-Fatigue score ranges from 0 to 52, with a higher score indicating less fatigue.
Visual Verbal Learning Test (VVLT) Score | Up to Day 2
  Assessment of cognition will be done by Visual Verbal Learning Test (VVLT) which includes 30 words in three consecutive word trials and the participants will be assessed for Immediate Recall and Delayed Recognition.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Leiden, Netherlands